CLINICAL TRIAL: NCT01261039
Title: Production of Vitamin D Metabolites by UV-radiation From Solar Bed
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Louise Lind Schierbeck, MD, research fellow, Hvidovre University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: h-3-2009-145
Record Dates: First submitted 2010-12-15; First posted 2010-12-16 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Production of Vitamin D in Skin When Exposed to UV-B by Solar Bed.
MeSH Terms: interventions — Ultraviolet Rays

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Solar bed UV-radiation (Active Comparator): Solar bed UV-radiation
  Interventions: Radiation: UV radiation
- Solar bed with UV filter (Sham Comparator): Solar bed with UV filter
  Interventions: Radiation: UV radiation

INTERVENTIONS:
Radiation: UV radiation — Subjects in both groups will be exposed to light in a solar bed for approximately 10 minutes (depending on Fitzpatrick skin type test) on the first day, but only one of the solar beds wields ultraviolet rays. The other has a filter, which filters out the ultraviolet rays.

SUMMARY:
Background:

Some patients do not readily absorb vitamin D from intestine. These patients may be helped by ultraviolet rays, which can come from sunlight or solar beds. When the skin is exposed to ultraviolet B rays (UVB) vitamin D is produced. This usually happens when the skin is exposed to sunlight. Vitamin D can also be ingested trough some foods, mainly fatty fish or supplements.

Vitamin D is important for bone, and long-term vitamin D deficiency can lead to osteoporosis. Vitamin D may also be important for the immune system-including autoimmune diseases-and the cardiovascular system.

Purpose:

The main purpose of the study is to learn more about the production of vitamin D3 in the skin, by ultraviolet radiation.

Study Course:

Day 0: Randomization. Subjects are randomized to two groups. Subjects in both groups will be exposed to light in a solar bed for approximately 10 minutes on the first day, but only one of the solar beds wields ultraviolet rays. The other has a filter, which filters out the ultraviolet rays.

Blood samples are drawn on the first day at following times: Before solar bed, after at 15 minutes, 1, 2, 4 and 6 hours.

Day 1,2,3 and 7 after solar bed exposure:

Blood samples are drawn and adverse events are registered.

ELIGIBILITY:
Inclusion Criteria:

Healthy adults

Exclusion Criteria:

Abnormal ALT or Creatinine Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-04; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Vitamin D 25-OHD | 8 days

SECONDARY OUTCOMES:
Changes in other calcium metabolic factors | 8 days
  Vitamin D3, Mg++, PTH, PO4--, Ca++

CONTACTS AND LOCATIONS:
Overall Officials: Jens-Erik B Jensen, MD, PhD, Study Chair — Hvidovre University Hospital; Louise L Schierbeck, MD, Study Chair — Dept. of Endocrinology; Ulrich Bang, MD, Study Chair — Hvidovre University Hospital; Jakob H Langdahl, Principal Investigator — University of Copenhagen
Locations (1):
- Hvidovre University Hospital, Hvidovre, Denmark

REFERENCES:
- [Derived] Langdahl JH, Schierbeck LL, Bang UC, Jensen JE. Changes in serum 25-hydroxyvitamin D and cholecalciferol after one whole-body exposure in a commercial tanning bed: a randomized study. Endocrine. 2012 Oct;42(2):430-5. doi: 10.1007/s12020-012-9641-z. Epub 2012 Mar 6. PMID 22391940